CLINICAL TRIAL: NCT00373191
Title: Effects of Surgery, Radiation Therapy, Chemotherapy, and Endocrine Therapy on High-Sensitivity C-Reactive Protein in Women With Operable Breast Cancer
Brief Title: Effect of Surgery, Radiation Therapy, Chemotherapy, and Hormone Therapy on Biomarkers in Women With Stage I, Stage II, Stage III Breast Cancer, or Ductal Carcinoma In Situ That Can Be Removed By Surgery
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: J0575 CDR0000485360; P30CA006973 (NIH); JHOC-J0575 (Other: SKCCC); JHOC-SKCCC-J0575 (Other: SKCCC)
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Drug Therapy; DNA Methylation; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum

INTERVENTIONS:
Drug: chemotherapy — N/A- not dictated by study
Drug: endocrine therapy — N/A- not dictated by study
Genetic: DNA methylation analysis — laboratory analysis
Genetic: protein analysis — laboratory analysis
Other: laboratory biomarker analysis — laboratory analysis
Other: questionnaire administration — questionnaire
Procedure: adjuvant therapy — N/A- not dictated by study
Procedure: conventional surgery — N/A- not dictated by study
Radiation: radiation therapy — N/A- not dictated by study

SUMMARY:
RATIONALE: Collecting and storing samples of blood from patients with cancer to study in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at the effects of surgery, radiation therapy, chemotherapy, and hormone therapy on biomarkers in women with stage I, stage II, stage III breast cancer, or ductal carcinoma in situ that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Measure the effects of surgery and radiation on concentrations of high-sensitivity C-reactive protein (hsCRP) in women with newly diagnosed stage I-III invasive breast cancer or ductal carcinoma in situ.
* Measure the effects of chemotherapy and/or endocrine therapy on concentrations of hsCRP in these patients.
* Summarize the differences in preoperative to peri-chemotherapy hsCRP concentrations separately for patients who do and who do not receive growth factors during chemotherapy.
* Observe the change in hsCRP concentrations and gene methylation over time with local and systemic treatment in these patients.
* Explore prevalence of baseline and change in methylation in a panel of genes that is known to be frequently and specifically hypermethylated in breast cancer.

OUTLINE: This is a prospective study.

A blood sample is collected at baseline, approximately 1 week after surgery, and at the time of a routine follow-up visit 3-6 months after completion of all local and systemic therapy, except for patients receiving endocrine therapy. For patients receiving adjuvant chemotherapy, a blood sample is collected prior to beginning chemotherapy and once during the final 2 courses of chemotherapy. For patients receiving radiotherapy, a blood sample is collected during the final 2 weeks of radiotherapy. For patients receiving endocrine therapy, a blood sample is collected between 2 and 6 months after starting endocrine therapy. Patients also complete a questionnaire about overall health and concurrent medications at baseline and during each follow-up visit.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically and/or cytologically confirmed stage I-III invasive breast carcinoma or ductal carcinoma in situ

  * Newly diagnosed disease
* Patient must be initiating a new course of treatment for breast carcinoma, including surgery (mastectomy or lumpectomy with or without nodal evaluation) with or without any of the following:

  * Radiation therapy
  * Chemotherapy
  * Endocrine therapy
* No known or suspected metastatic disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* No infectious or inflammatory condition, at the discretion of the principal investigator
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

* More than 6 months since prior surgery

  * Fine-needle aspirate or biopsy allowed
* More than 6 months since prior radiotherapy
* More than 6 months since prior chemotherapy
* More than 6 months since prior endocrine therapy
* No neoadjuvant endocrine therapy or chemotherapy
* More than 2 weeks since prior and no concurrent regular use of any of the following:

  * Hydroxymethyl glutaryl coenzyme A reductase inhibitor (statin)
  * Nonsteroidal anti-inflammatory drug (NSAID)*
  * Cyclooxygenase-2 (COX-2) inhibitor
  * Aspirin*
* Acetaminophen and opioid use is permitted as needed NOTE: *Use of these products ≤ 2 times per week at standard over-the-counter doses allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed ductal carcinoma in situ or invastive breast cancer.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2006-05; Primary Completion 2009-02 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in high-sensitivity C-reactive protein and gene methylation over time | indefinite

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States